CLINICAL TRIAL: NCT03797612
Title: A Phase 2 Randomized Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a Single Intrathecal Preoperative Administration of Brivoligide Injection in Patients With a Pain Catastrophizing Scale Score ≥16 Undergoing Unilateral Total Knee Arthroplasty
Brief Title: Study to Evaluate a Preop Dose of Brivoligide Injection for Pain After Knee Replacement in Patients With High PCS Scores
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study initiation delayed due to COVID 19
Sponsor: Adynxx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADYX-005
Record Dates: First submitted 2019-01-06; First posted 2019-01-09 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Pain, Postoperative
Keywords: Knee replacement; TKA; Total Knee Arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brivoligide Injection 660 mg/6 mL (Experimental): Subjects randomized to the active treatment group will receive a single 660 mg/6 mL intrathecal administration of brivoligide injection as a slow bolus injection just prior to administration of spinal anesthesia, via the same needle.
  Interventions: Drug: Brivoligide Injection 660 mg/6 mL
- Placebo 6 mL (Placebo Comparator): Subjects randomized to the placebo group will receive a single 6 mL intrathecal injection of placebo as a slow bolus injection just prior to administration of spinal anesthesia, via the same needle.
  Interventions: Drug: Placebo 6 mL

INTERVENTIONS:
Drug: Brivoligide Injection 660 mg/6 mL — Single preoperative intrathecal injection
  Other Names: AYX1 Injection 660 mg/6 mL
  Arms: Brivoligide Injection 660 mg/6 mL
Drug: Placebo 6 mL — Single preoperative intrathecal injection
  Arms: Placebo 6 mL

SUMMARY:
This is a multi-center, Phase 2, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of brivoligide injection administered intrathecally before surgery in patients with a Pain Catastrophizing Scale (PCS) score ≥16 undergoing primary unilateral total knee arthroplasty.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and postoperative pain reducing efficacy of a single preoperative intrathecal administration of brivoligide injection in patients with a Pain Catastrophizing Scale (PCS) score ≥16 undergoing unilateral total knee arthroplasty.

Potential subjects will be prescreened for PCS scores of 16 or greater in advance; pre-qualified patients will be invited to the investigative site for informed consent and full screening within 30 days of randomization. Patients providing informed consent and meeting all study eligibility criteria will be enrolled in the study on the day of surgery (Day 1). Safety assessments will be performed through Day 28; efficacy assessments will be conducted at the follow-up visits and daily via electronic diary by subjects through Day 42. Follow up visits will occur on Days 7, 14, 21, 28, and 42.

ELIGIBILITY:
Inclusion Criteria:

* Score of 16 or greater on the PCS scale
* Scheduled for primary unilateral TKA with spinal anesthesia as the primary anesthetic for painful osteoarthritis without congenital knee pathology
* American Society of Anesthesiologists Physical Status Classification System ≤ 3
* Medically stable for elective surgery with spinal anesthetic as determined by the Investigator
* Body mass index of 18-45 kg/m2
* Stable medical regimen at least 1 week before randomization
* Able to read and understand study instructions in English or Spanish, and willing to comply with all study procedures

Exclusion Criteria:

* Target knee > 20 degrees valgus or varus deformity, evidence of significant bone loss or ligamentous laxity, or existing major hardware that requires removal during TKA
* Inflammatory arthridities (e.g., rheumatoid arthritis, lupus, ankylosing spondylitis, psoriatic arthritis), with the exception of clinically stable/non-active gout
* Undergoing concomitant surgical procedures or non-elective TKA, or contralateral knee is likely to require TKA within 6 weeks (or would interfere with study assessments)
* Use of cryoneurolysis (including Iovera) on the current operative knee region within 6 months prior to randomization and/or at any time through the duration of the study
* Planned use of general anesthesia as the primary anesthetic; planned use of neuroaxial (intrathecal or epidural) opioids, or any use of extended release/long acting opioids or ketamine preoperatively and/or at any time through the duration of the study
* Use of more than 40 mg per day (on average) of oral morphine or its equivalent within 1 month prior to randomization
* Current neurologic disorder, which could confound the assessment of pain (e.g., Parkinson's, Multiple Sclerosis)
* Unstable mental condition and/or evidence of an uncooperative attitude in the opinion of the Investigator; subjects diagnosed with schizophrenia, prescribed antipsychotic medications or MAOIs
* Women who are pregnant or nursing
* Subjects engaged in pending or active litigation, or seeking disability compensation; subjects whose cases have been settled or finally decided are not excluded
* Participation in a clinical trial with the last dose or intervention within 1 month of randomization, or planned participation in a clinical trial during this study
* Previous participation in any study involving brivoligide injection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) Pain with Walking 15 Meters | Day 7 to Day 28
  Least squares mean pain rating (NRS) with walking during the 15-meter walk Day 7 to Day 28

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) Pain at Rest | Day 7 to Day 28
  Least squares mean pain rating (NRS) at rest Day 7 to Day 28
Numerical Rating Scale (NRS) Pain with 90 Degrees Passive Knee Flexion | Day 7 to Day 28
  Least squares mean pain rating (NRS) with passive knee flexion to 90 degrees from Day 7 to Day 28
Total Postoperative Opioid Use | Postoperative through Day 42
  Total use of postoperative opioid medications (morphine equivalents) to Day 42
Time to Numerical Rating Scale (NRS) Pain ≤ 3 for Worst Pain | Postoperative through Day 42
  Time to achieve NRS pain score ≤ 3 for worst pain

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Sheffield, Alabama
  - Research Site, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.